CLINICAL TRIAL: NCT00975936
Title: A Human Phase 0, Microdose Drug-Drug Interaction Study With [14C]-GSK706769 and Ketoconazole in Healthy Male Volunteers
Brief Title: Phase 0 Microdose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 113191
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Autoimmune Diseases
Keywords: Microdose; Drug-Drug Interaction; Ketoconazole; Phase 0
MeSH Terms: conditions — Autoimmune Diseases | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- [14C]-GSK706769 (Experimental): Single dose of 50µg [14C]-GSK706769 containing 250 nCi
  Interventions: Drug: [14C]-GSK706769
- [14C]-GSK706769 + Ketoconazole (Experimental): An oral, 5-day repeat dose of 200 mg Ketoconazole (Q12) with a concomitant single oral dose of 50 µg [14C]-GSK706769 containing 250 nCi on day 3.
  Interventions: Drug: [14C]-GSK706769; Drug: Ketoconazole

INTERVENTIONS:
Drug: [14C]-GSK706769 — 50µg [14C]-GSK706769 containing 250 nCi
Drug: Ketoconazole — 200 mg Ketoconazole (Q12)
  Arms: [14C]-GSK706769 + Ketoconazole

SUMMARY:
This study is a methodology study to evaluate a microdose strategy for Drug-Drug Interaction (DDI) which will be useful in the evaluation of the backup compounds for GSK706769, as well as possibly other assets. The safety, tolerability and pharmacokinetics will be evaluated in healthy adult subjects. This will be an open-label fixed-sequence 2-period study in healthy male volunteers after oral administration of [14C]-GSK706769 alone and in the presence of Ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-50 years of age inclusive, at the time of signing the informed consent.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Signed written informed consent prior to beginning study-related procedures. Subjects must understand the aims, investigational procedures and possible consequences of the study and must be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 7 days post-last dose.
* Body weight greater than or equal to 50 kg (110 pounds) and body mass index (BMI) between 19 and 35 kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined in the protocol.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications (including Ketoconazole), or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Any medical or surgical conditions that might significantly interfere with the gastrointestinal absorption, distribution, metabolism, or excretion of the study drugs (eg, gastrectomy).
* Subjects who have been involved in a 14C human research study within the previous 12 months.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication until the completion of the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2009-11-12 (Actual); Study Completion 2009-11-12 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC0-t. AUC0-infinity, total plasma clearance (CL/F), apparent volume of distribution (V/F) and terminal phase half-life (t1/2) will also be calculated where data permit. | Throughout study

SECONDARY OUTCOMES:
Clinical safety and tolerability data including spontaneous Adverse Event reporting, ECGs, vital signs, nursing/physician observation, physical examination and clinical laboratory values. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States

REFERENCES:
- See also: Results for study 113191 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113191?search=study&search_terms=113191#rs